CLINICAL TRIAL: NCT00000423
Title: Social Support and Health in Fibromyalgia
Brief Title: Support, Health, and Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: R01AR044020 (NIH); R01AR044020 (NIH); NIAMS-029
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-03

CONDITIONS: Fibromyalgia; Quality of Life
Keywords: Fibromyalgia; Health education; Program evaluation; Social support; Managed care; Quality of well-being
MeSH Terms: conditions — Fibromyalgia; Health Education | interventions — Self-Help Groups

INTERVENTIONS:
Behavioral: Social support group
Behavioral: Social support and education group

SUMMARY:
This study tests the effects of social support and education on the health and well-being of people with fibromyalgia (FMS). We recruited 600 adults with a confirmed diagnosis of FMS from a large health maintenance organization. We randomly assigned the study participants to one of three groups. People in the social support group met with others who suffer from FMS for 2 hours every week for 10 weeks, and then monthly for an additional 10 months. The social support and education group also had 10 2-hour weekly meetings followed by 10 monthly meetings with others who suffer from FMS. Members of this group learned about the disease and ways they can manage it themselves. The third group participated only in the five assessment periods. The study lasted 4 years.

DETAILED DESCRIPTION:
Next to osteoarthritis, FMS is the most common arthritis-related disease. Symptoms include musculoskeletal pain, fatigue, headaches, irritable bowel syndrome, morning stiffness, and sleep disturbances. Fluctuating severity, pain, and frustration with the difficulty of diagnosis and treatment lead patients to continually seek help from health care professionals. There is no known cause or cure for this disease.

This study tests the effects of social support and education on the health and well-being of people with fibromyalgia (FMS). We recruited 600 adults with a confirmed diagnosis of FMS from a large health maintenance organization. To be eligible, people had to meet the American College of Rheumatology guidelines for FMS. After we confirmed the diagnosis, we assigned those who agreed to participate to one of three groups. The first group (social support) met with others who suffer from FMS for 2 hours every week for 10 weeks, and then monthly for an additional 10 months. The second group (social support and education) also had 10 2-hour weekly meetings followed by 10 monthly meetings with others who suffer from FMS, and its members learned about the disease and self-management techniques. The third group (control) participated only in the five assessment periods. We assessed people in all three groups before we assigned them to a group, after the intervention, and at yearly follow-ups. The study duration was 4 years.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of fibromyalgia documented in medical records and confirmed using The American College of Rheumatology criteria for classification of FMS: (1) A history of widespread pain (pain on both sides of the body, above and below the waist, and present for at least 3 months). (2) Pain in 11 or more of 18 tender-point sites.
* Patient willing to attend 10 weekly meetings and 10 monthly meetings.

Exclusion Criteria:

* Patients who do not meet ACR criteria for FMS described above.
* Patients who cannot attend meetings once a week for 10 weeks and once a month for 10 months were excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 1996-09; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Overall Officials: Thereasa A. Cronan, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

REFERENCES:
- [Result] Oliver K, Cronan TA, Walen HR, Tomita M. Effects of social support and education on health care costs for patients with fibromyalgia. J Rheumatol. 2001 Dec;28(12):2711-9. PMID 11764222